CLINICAL TRIAL: NCT03804502
Title: Pilot Study of TearCare System - Long-Term Extension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06215
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TearCare (Experimental): Subjects will receive one TearCare treatment at the baseline visit
  Interventions: Device: TearCare

INTERVENTIONS:
Device: TearCare — The TearCare System warms the eyelids to melt the meibum by applying heat to the external surface of the eyelids for 15 minutes. Following completion of the thermal portion of the procedure, the clinician performs manual expression of each of the eyelids.

SUMMARY:
The objective of the study is to evaluate the long-term clinical utility, safety, and effectiveness of re-treatment with the TearCare™ System in adult patients with dry eye syndrome who had previously been treated with the TearCare System.

DETAILED DESCRIPTION:
This was an extension of an initial 6-month, prospective, single-center, randomized, parallel-group pilot study (NCT03006978). In the initial study, subjects with dry eye disease (DED) were randomized to either a single TearCare® treatment or 4 weeks of daily warm compress therapy. The extension study involved retreatment of those subjects assigned to the TearCare® treatment group following the initial 6-month end point. At 6 months, subjects were evaluated for the clinical signs and symptoms of DED prior to retreatment in the extension study that would measure the safety, effectiveness, and durability of a TearCare® retreatment for another 6 months through a 12-month end point.

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled in the TearCare arm of the TearCare Pilot Study
* Reports dry eye symptoms within 3 months of the baseline examination with a Standard Patient Evaluation for Dryness (SPEED) score ≥ 6
* TBUT of <10 seconds in at least one eye
* Willing to comply with the study, procedures, and follow-up
* Willing and able to provide consent

Exclusion Criteria:

* Any active ocular or peri-ocular infection or inflammation
* Recurrent eye inflammation within the past 3 months
* Ocular surgery, oculoplastic surgery, ocular injury, Ocular Herpes Simplex, or Herpes Zoster
* Ocular surface abnormalities that may affect tear film distribution or treatment
* Abnormal eyelid function in either eye
* Diminished or abnormal facial, periocular, ocular or corneal sensation
* Ocular surface abnormalities such as corneal epithelial defects, ulcers, corneal dystrophies
* Systemic diseases resulting in dry eye (e.g. Sjogren's syndrome)
* Allergies to silicone tissue adhesives
* An absence or fibrosis of the Meibomian glands (e.g. ectodermal dysplasia).
* Unwillingness to abstain for the duration of the study from systemic medication known to cause ocular dryness (e.g. Accutane, antihistamines, etc.)
* Anyone who requires chronic use (i.e. for any portion of the study) of topical ophthalmic antibiotics, steroids, non-steroidal anti-inflammatory medications or who has been on any of these medications within the past 30 days.
* Unwillingness to washout and remain off certain dry eye medications for the duration of the study.
* Participation in another ophthalmic clinical trial within the past 30 days
* Co-existing conditions that could interfere with the assessment of safety or efficacy of treatment (e.g. macular disease, pregnancy, nursing, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Badawi, MD, Principal Investigator — Sight Sciences, Inc.
Locations (1):
- Central Eye Care, Arlington Heights, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TearCare
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Arm/Group | TearCare
Number analyzed (Participants) | 12
Number analyzed (eyes) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Tear Break Up Time [Mean (Standard Deviation); unit: seconds] — The TBUT was evaluated by measuring the time to breakup of the tear film following a complete blink when viewed through the slit-lamp using a cobalt blue filter. The TBUT was recorded using a stopwatch for each eye as the average of 3 measurements at each visit. The TBUT value for both eyes of a subject was then averaged resulting in a single TBUT value for each subject
  seconds | 5.0 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Tear Break-Up Time From Extension Study Baseline to Month 1
Description: The TBUT was evaluated by measuring the time to breakup of the tear film following a complete blink when viewed through the slit-lamp using a cobalt blue filter. The TBUT was recorded using a stopwatch for each eye as the average of 3 measurements at each visit. The change in TBUT was The difference between the mean baseline value and the mean Month 1 value. The TBUT for each eye for a subject was averaged resulting in a single TBUT value for each subject (n=12).
Time Frame: 1 month
Population: All subjects that had been randomized to TearCare in the initial pilot study (NCT03006978) and consented to participate in the extension study.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | TearCare
Number analyzed (Participants) | 12
Number analyzed (eyes) | 24
seconds | 12.4 (3.3)

2. Secondary Outcome: Mean Change in Meibomian Gland Score From Extension Study Baseline to Month 1
Description: Using a Korb Meibomian Gland Evaluator (TearScience), the meibomian gland assessment was conducted by evaluating the consistency of the secretions that were observed upon expression of meibomian glands in the nasal, central, and temporal regions of the lower eyelids. The central, consecutive 5 glands in each region were evaluated. The instrument was held at the eyelid margin for 10-15 seconds, and the secretions were graded on a 0-3 scale for each gland (0=no expression; 1=toothpaste; 2=cloudy; and 3=clear), with a 0 (worst)-45 (best) score range for each eye. The score for each eye of a subject was averaged. The change from baseline in the Meibomian Gland Score is the difference between the mean baseline value and the mean value at Month 1. A positive value for change is an improvement
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | TearCare
Number analyzed (Participants) | 12
Number analyzed (eyes) | 24
units on a scale | 19.5 (8.4)

3. Secondary Outcome: Mean Change in SPEED II Questionnaire Result From Extension Study Baseline to Month 1
Description: The Standard Patient Evaluation for Eye Dryness II (SPEED II) questionnaire is a well-validated instrument and widely used assessment tool for dry eye indications. The SPEED II questionnaire was used to evaluate the symptoms of study subjects. The SPEED II survey measures the severity (0-4 scale) and frequency (0-3 scale) of DED symptoms. The SPEED score was calculated by adding the total of the frequency and severity scores; a score of greater than or equal to 6 may be an indicator of DED (range 0 [best] to 7 [worst]). The reported value is the mean of the change for all subjects. A negative result indicates improvement.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TearCare
Number analyzed (Participants) | 12
units on a scale | -2.9 (2.7)

4. Secondary Outcome: Mean Change in OSDI Questionnaire Result From Extension Study Baseline to Month 1.
Description: The Ocular Surface Disease Index (OSDI) is a 12-item questionnaire that assesses symptoms of ocular irritation associated with dry eye and the impact of these on vision-related activities. The OSDI score ranges from 0 (best possible) to 100 (worst possible). The change in OSDI questionnaire from baseline to Month 1 is the difference between the scores at the two timepoints. A negative value would indicate improvement and a positive value, a worsening. The reported value is the mean of the change for all subjects.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TearCare
Number analyzed (Participants) | 12
units on a scale | -11.2 (14.8)

5. Secondary Outcome: Mean Change in Corneal Staining From Extension Study Baseline to Month 1
Description: Corneal (fluorescein) staining scores was recorded to assess the integrity of the ocular surface. The severity of staining was assessed and quantified using the National Eye Institute/Industry Grading System scoring 5 regions of the cornea using a scale from 0 to 3 (normal-severe) for each region. The scores for the regions of the cornea were added to obtain a total score that ranged from 0 (best) to 15 (worst). The score for each eye of a subject was averaged. The mean change from baseline to month 1 is the difference in the two scores. A negative result indicates improvement.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | TearCare
Number analyzed (Participants) | 12
Number analyzed (eyes) | 24
units on a scale | -0.17 (.33)

6. Secondary Outcome: Mean Change in Conjunctival Staining From Extension Study Baseline to Month 1
Description: Conjunctival (lissamine green) staining scores was recorded to assess the integrity of the ocular surface. The severity of staining was assessed and quantified using the National Eye Institute/Industry Grading System scoring 6 regions of the conjunctiva using a scale from 0 to 3 (normal-severe) for each region. The scores for the regions of the conjunctiva were added to obtain a total score that ranged from 0 (best) to 18 (worst). The score for each eye of a subject was averaged. The mean change from baseline to month 1 is the difference in the two scores. A negative result indicates improvement.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | TearCare
Number analyzed (Participants) | 12
Number analyzed (eyes) | 24
units on a scale | -0.54 (1.25)

7. Secondary Outcome: Mean Change in SANDE Result From Extension Study Baseline to Month 1
Description: The SANDE (Symptom Assessment iN Dry Eye) instrument is a simple 2-item questionnaire, that focuses on the frequency and the severity of dry eye symptoms with each measured along a visual analog scale. SANDE, because of its simplicity, is often used in routine clinical practice. For the core questions, the frequency and severity scores are multiplied together, and the square root is taken to produce an overall SANDE score from 0 (best possible) to 100 (worst possible). The mean change from baseline to month 1 is the difference in the two scores. A negative result indicates improvement.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TearCare
Number analyzed (Participants) | 12
score on a scale | -13.2 (15.6)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | TearCare
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TearCare (N=8)
mild allergic conjunctivitis (General disorders) | 1 (1) — non-ocular

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT03804502/Prot_SAP_000.pdf